CLINICAL TRIAL: NCT03459261
Title: Can we Improve the Treatment of Acute Posttraumatic Osteomyelitis in Patients With High-energy Tibial Fractures by Using Perioperative Immunoinflammatory Markers?
Brief Title: Acute Posttraumatic Osteomyelitis in Patients With High-energy Tibial Fractures and Biomarkers
Acronym: POMTIBIAL
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Prof. Alojz Ihan, MD, Ph.D, Institute of Microbiology and Immunology, Ljubljana, Slovenia (Unknown)
Responsible Party: Principal Investigator, Matjaž Groznik, MD, Head of HDU at Traumatology Department Matjaž Groznik, MD, Specialist in Traumatology and Intensive Care Medicine, University Medical Centre Ljubljana
Other Study IDs: 20120130
Record Dates: First submitted 2018-02-10; First posted 2018-03-08 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Osteomyelitis Tibia; Surgical Site Infection
Keywords: osteomyelitis; tibial fracture; cytokines; PCT; CRP; albumin
MeSH Terms: conditions — Surgical Wound Infection; Osteomyelitis; Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POM: post-traumatic osteomyelitis group (POM), the participants who developed post-traumatic osteomyelitis after primary surgical treatment and were taken blood sample on admission (ADD), first postoperative day (POD1) and fourth postoperative day (POD4). Patients were included in POM group after additional assessment of meeting the CDC/NHSN surveillance definition criteria for osteomyelitis: positive intraoperative withdrawal bone and soft tissue sample, types of cultured bacteria, histopathologic proof of osteomyelitis and clinical signs of surgical site infection.
  Interventions: Diagnostic Test: blood sample on admission (ADD), first postoperative day (POD1) and fourth postoperative day (POD4)
- NO POM: No POM group, the participants who did not develop postraumatic osteomyelitis to tibia after primary surgical treatment and were taken blood sample on admission (ADD), first postoperative day (POD1) and fourth postoperative day (POD4) in follow up interval of 6 months /control group/. Patients were included in No POM group after assessment of not meeting the CDC/NHSN surveillance definition criteria for osteomyelitis.

INTERVENTIONS:
Diagnostic Test: blood sample on admission (ADD), first postoperative day (POD1) and fourth postoperative day (POD4) — Laboratory analyses of peripheral venous blood on admission (blood sample ADD), 24 hours after surgery (blood sample POD1) and fourth-day after surgery (blood sample POD4) included biochemical analysis, complete blood count, C-reactive protein (CPR), procalcitonin (PCT), albumin/protein level, prothrombin time and international normalized ratio (INR) (only on admission) and for determination of cytokines: tumor necrosis factor alpha (TFN-α), interleukin-6 (IL-6), interleukin-10 (IL-10).
  Groups: POM

SUMMARY:
The present trial was aimed to identify which biomarkers could be associated in perioperative period after surgical treatment of tibial fracture to the development of POM.

DETAILED DESCRIPTION:
Early diagnosis of acute posttraumatic osteomyelitis (POM) is of vital importance for avoiding devastating complications. Diagnosing POM is difficult due to the lack of a highly specific and sensitive test, such as in myocardial infarct, stroke and intracranial bleeding. Serum inflammatory markers, C-reactive protein (CRP), procalcitonin (PCT), white blood cells (WBC) can support clinical findings but they are not able to differentiate between inflammatory response to infection and the host response to non-infection insult with high specificity and sensitivity.

The prospective nonrandomised cohort study included 86 patients after high-energy injury to the shin requiring primary surgical treatment (open or closed reduction and internal fixation of tibial fracture). Values of the biochemical and immunoinflammatory profile were measured on admission (ADD), first postoperative day (POD1) and fourth-postoperative day (POD4).

The objectives of the study were to investigate that the biochemical and immunoinflammatory profile could facilitate postoperative monitoring, guide the antibiotic treatment and timing of revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* high-energy injury to proximal, shaft or distal tibia,
* tibial fracture requiring primary surgical treatment /ORIF

Exclusion Criteria:

* ankle fracture,
* patella fracture,
* avulsion fracture of the knee,
* malignant neoplasm and pathological tibial fracture,
* systemic autoimmune disease of connective tissue,
* immature patients under 15 years of age (children),
* immunocompromised patients.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Department of Traumatology at University Clinical Centre Ljubljana were included after written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Measurement of biomarkers CRP, PCT, WBC on ADD, POD1, POD4 | perioperative period
  WBC count (reference range 4-10 x 109/L), WBC differential (neutrophil count 1.50-7.40 x 109/L, lymphocyte count 1.10-3.50 x 109/L) and hematocrit (reference range 0.390-0.500) were analyzed with a hematological blood analyzer LH75 (Beckman Coulter). The immunocytochemic analyzer Modular Analytics SWE (Roche Diagnostics) was used for serum samples analysis. The serum concentration of CRP (reference range 0-5mg/L) was measured by the immunoturbidimetric method, PCT (reference range 0-0.5μg/L) by the electrochemiluminescence method and albumins (reference range 35-52g/L) by the bromcresol green method.
Assessment of patients' immune status | perioperative period
  Whole venous blood was collected into vacutainer tubes containing EDTA. Samples were processed for flow cytometry. For surface staining, the standard whole-blood staining methodology as prescribed by the manufacturer (BDBiosciences) was used. For detecting regulatory T cells, samples were stained for surface antigens with a mix of anti-CD25-PE/ anti-CD127-APC/ anti-CD4-PE-Cy™7. All antibodies were obtained from BDBiosciences (Mountain View, Ca, USA). Cells were analyzed on FACSCantoII™ Flow Cytometer (BDBiosciences) equipped with blue (488-nm solid-state) and red (633-nm helium-neon) laser. Digital data was acquired with FACSDiva software (BDBiosciences) and analyzed using FlowJo software (Tree Star Inc.,).
Determination of cytokines level in serum: tumor necrosis factor (TFN-alpha), interleukin-6 (IL-6), interleukin-10 (IL-1) and lymphocyte populations | perioperative period
  Cytokine concentrations were measured by commercially available enzyme-linked immunosorbent assay (ELISA) kits. TNF-α (Milenia Biotec, Germany), IL-6 and IL-10 (Thermo Scientific, USA) were measured according to the manufacturer's instructions.